CLINICAL TRIAL: NCT06830109
Title: Nasal Obstruction Randomized Trial With Oxymetazoline and Corticosteroids
Brief Title: Nasal Obstruction With Oxymetazoline and Corticosteroids
Acronym: NORTOC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Nyssa Farrell, Assistant Professor of Otolaryngology-Head & Neck Surgery, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202406175
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Nasal Obstruction
Keywords: Oxymetazoline; Corticosteroids; Chronic rhinitis
MeSH Terms: conditions — Nasal Obstruction | interventions — Oxymetazoline; Budesonide

STUDY DESIGN:
Intervention Model Description: Single-center, double-blinded, randomized, controlled trial conducted at Washington University School of Medicine
Who Masked: Participant, Investigator
Masking Description: The participant and the research team will be unaware of the participant's intervention assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- budesonide + oxymetazoline, (Experimental): alpha-adrenergic agonist and vasoconstrictor that is available over-the-counter (OTC).
  Interventions: Drug: Oxymetazoline Nasal Spray; Drug: Budesonide nasal spray
- budesonide (Active Comparator): intranasal corticosteroid that is available OTC.
  Interventions: Drug: Budesonide nasal spray

INTERVENTIONS:
Drug: Oxymetazoline Nasal Spray — Intra-nasal alpha-adrenergic agonist and vasoconstrictor that is available over-the-counter (OTC)
  Other Names: Afrin (commercial name for oxymetazoline hydrochloride)
  Arms: budesonide + oxymetazoline,
Drug: Budesonide nasal spray — Intranasal corticosteroid that is available over-the-counter (OTC)
  Other Names: Rhinocort (commercial name for budesonide)

SUMMARY:
This study aims to examine the efficacy and safety of commination oxymetazoline/intranasal steroids for long-term management of chronic nasal obstruction that is recalcitrant to the current standard of care. The investigators hypothesize that combination treatment with oxymetazoline and intranasal corticosteroid spray will provide a larger reduction in nasal obstruction than intranasal corticosteroid alone for patients suffering from chronic nasal obstruction, and there will not be occurrences of rhinitis medicamentosa.

DETAILED DESCRIPTION:
Participants will be directed to apply the intranasal spray, at a dosage of two sprays in each nostril, twice daily. The total treatment time for participants in both trial arms is 7 weeks. Participants will be randomized to either 1) oxymetazoline + budesonide intranasal spray or 2) budesonide intranasal spray. Participants will be mailed the intranasal spray directly from the pharmacy. Participants will complete questionnaires via REDCap survey link at baseline, Week 2, Week 4, Week 5, Week 6, and Week 7. A group of 10 participants will be asked to have nasal mucosal biopsies done at baseline and between weeks 4 and 6.

ELIGIBILITY:
Inclusion Criteria:

1. males and females ages 18 years or older
2. have a history of nasal obstruction
3. have failed a trial of topical steroids (that included at least 1 month of daily use)
4. ability to read, write, and understand English
5. either do not desire surgery or are poor surgical candidates due to medical comorbidities.
6. Patients who have had prior use of oxymetazoline or other nasal decongestants are eligible for the study but must have stopped usage 4 weeks prior to randomization.

   1. Must be willing to stop using any other nasal sprays, besides saline, and oral decongestants.

Exclusion Criteria:

1. Any history of sinonasal mass/tumor
2. Any history of nasal polyps
3. a known history of chronic sinusitis
4. an allergy to oxymetazoline
5. or who have any medical contraindication to oxymetazoline use, such as pulmonary hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-10-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Responders | 4 weeks
  The primary outcome measure will be the rate of responders (as a percentage) to the intervention defined as the number of participants reporting 2 (Moderately Improved), or 3 (Much Improved) in the Clinical Global Impression of Improvement (CGI-I) assessed after 4 weeks of treatment divided by the total number of participants in each study group.
  CGI-I asks subjects to rate their overall response to treatment using a 7-point Likert scale ranging from -3 to 3 ("Much Worse" to "Much Improved"). Participants responding 2 (Moderately Improved), or 3 (Much Improved) to the the CGI-I question "Compared to the start of the study, how would you rate your nasal breathing now", will be defined as responders to treatment.

SECONDARY OUTCOMES:
Sino-Nasal Outcome Test (SNOT-22) | baseline, 2 weeks, and 4 weeks
  SNOT-22 is a 22-question survey designed to measure the physical, functional, and emotional consequences of rhinosinusitis. It contains questions regarding symptoms commonly associated with sinonasal disease.
  Subjects rate each question by using a 0-5 point scale with 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The SNOT-22 total score ranges from a minimum score of 0 to a maximum score of 110, with higher scores representing worse outcome.
Nasal Obstruction Symptom Evaluation (NOSE) | baseline, 2 weeks, 4 weeks
  NOSE is a disease-specific survey designed to measure nasal obstruction. It consists of 5 questions, each rated on a scale of 0 to 4. The total score represents the sum of the raw scores multiplied by 5 and ranges from 0 to 100, with higher values indicating worse symptoms. A score of 30 is considered indicative of clinically significant nasal airway obstruction.
Clinical Global Impression of Severity (CGI-S) | baseline, week 4
  The CGI-Severity Scale from 1 to 7 (1 is "Not Obstructed at All", 7 is "Completely Obstructed") provides the severity of nasal obstruction as perceived from the patient. Comparison of CGI-S scores at 4 weeks with baseline will help identify subjects that have experienced rebound congestion. The investigators will report the number of patients who report a worsening of their symptoms, as measured by a 1-point (1 category) increase in CGI-S scale at 4 weeks as compared to CGI-S scale at baseline.

OTHER OUTCOMES:
Clinical Global Impression of Severity (CGI-S); experimental arm | baseline, week 7
  The CGI-Severity Scale from 1 to 7 (1 is "Not Obstructed at All", 7 is "Completely Obstructed") provides the severity of nasal obstruction as perceived from the patient. Comparison of CGI-S scores at 7 weeks with baseline will help identify subjects in the experimental arm who struggled with discontinuation of oxymetazoline. The investigators will report the number of subjects who report a worsening of their symptoms, as measured by a 2-point (2 categories) increase in CGI-S scale at 7 weeks as compared to CGI-S scale at baseline in the experimental arm only.

CONTACTS AND LOCATIONS:
Overall Officials: Nyssa F Farrell, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scarupa MD, Kaliner MA. Nonallergic rhinitis, with a focus on vasomotor rhinitis: clinical importance, differential diagnosis, and effective treatment recommendations. World Allergy Organ J. 2009 Mar;2(3):20-5. doi: 10.1097/WOX.0b013e3181990aac. PMID 23282951
- [Background] Stewart M, Ferguson B, Fromer L. Epidemiology and burden of nasal congestion. Int J Gen Med. 2010 Apr 8;3:37-45. doi: 10.2147/ijgm.s8077. PMID 20463822
- [Background] Thongngarm T, Assanasen P, Pradubpongsa P, Tantilipikorn P. The effectiveness of oxymetazoline plus intranasal steroid in the treatment of chronic rhinitis: A randomised controlled trial. Asian Pac J Allergy Immunol. 2016 Mar;34(1):30-7. doi: 10.12932/AP0649.34.1.2016. PMID 26994623
- [Background] Calvo-Henriquez C, Viera-Artiles J, Rodriguez-Iglesias M, Rodriguez-Rivas P, Maniaci A, Yanez MM, Martinez-Capoccioni G, Alobid I. The Role of Corticosteroid Nasal Irrigations in the Management of Chronic Rhinosinusitis: A State-of-the-Art Systematic Review. J Clin Med. 2023 May 22;12(10):3605. doi: 10.3390/jcm12103605. PMID 37240711
- [Background] Vaidyanathan S, Williamson P, Clearie K, Khan F, Lipworth B. Fluticasone reverses oxymetazoline-induced tachyphylaxis of response and rebound congestion. Am J Respir Crit Care Med. 2010 Jul 1;182(1):19-24. doi: 10.1164/rccm.200911-1701OC. Epub 2010 Mar 4. PMID 20203244
- [Background] Graf P, Juto JE. Decongestion effect and rebound swelling of the nasal mucosa during 4-week use of oxymetazoline. ORL J Otorhinolaryngol Relat Spec. 1994 May-Jun;56(3):157-60. doi: 10.1159/000276633. PMID 7515487
- [Background] Morris S, Eccles R, Martez SJ, Riker DK, Witek TJ. An evaluation of nasal response following different treatment regimes of oxymetazoline with reference to rebound congestion. Am J Rhinol. 1997 Mar-Apr;11(2):109-15. doi: 10.2500/105065897782537197. PMID 9129752
- [Background] Kumar RS, Jain MK, Kushwaha JS, Patil S, Patil V, Ghatak S, Sanmukhani J, Mittal R. Efficacy and Safety of Fluticasone Furoate and Oxymetazoline Nasal Spray: A Novel First Fixed Dose Combination for the Management of Allergic Rhinitis with Nasal Congestion. J Asthma Allergy. 2022 Jun 10;15:783-792. doi: 10.2147/JAA.S357288. eCollection 2022. PMID 35712651
- [Background] Matreja PS, Gupta V, Kaur J, Singh S. Efficacy of fluticasone and oxymetazoline as the treatment for allergic rhinitis. J Clin Diagn Res. 2012;6(1):85-88.
- [Background] Meltzer EO, Bernstein DI, Prenner BM, Berger WE, Shekar T, Teper AA. Mometasone furoate nasal spray plus oxymetazoline nasal spray: short-term efficacy and safety in seasonal allergic rhinitis. Am J Rhinol Allergy. 2013 Mar-Apr;27(2):102-8. doi: 10.2500/ajra.2013.27.3864. PMID 23562197
- [Background] Juvekar MR, Vaidya GK, Majumder A, Pendharkar AD, Irudhayarajan A, Kundu A, Ramesh D, Kumar JD, Jagannatha B, Mathew J, Nikam MP, Mehta M, Chawla N, Hajare P, Gowda PGC, Murthy PVLN, Mathew SM, Damle MV, Kant C, Nair AB, Jaiswal A, Mehta RT. A Real-World Observational Study to Evaluate the Safety and Effectiveness of Fluticasone Furoate-Oxymetazoline Fixed Dose Combination Nasal Spray in Patients with Allergic Rhinitis. Clin Drug Investig. 2024 Feb;44(2):123-130. doi: 10.1007/s40261-023-01338-8. Epub 2024 Jan 9. PMID 38195833
- [Background] Elwany SS, Stephanos WM. Rhinitis medicamentosa. An experimental histopathological and histochemical study. ORL J Otorhinolaryngol Relat Spec. 1983;45(4):187-94. doi: 10.1159/000275642. PMID 6192384
- [Background] Elwany S, Abdel-Salaam S. Treatment of rhinitis medicamentosa with fluticasone propionate--an experimental study. Eur Arch Otorhinolaryngol. 2001 Mar;258(3):116-9. doi: 10.1007/s004050000309. PMID 11374251
- [Background] Knipping S, Holzhausen HJ, Goetze G, Riederer A, Bloching MB. Rhinitis medicamentosa: electron microscopic changes of human nasal mucosa. Otolaryngol Head Neck Surg. 2007 Jan;136(1):57-61. doi: 10.1016/j.otohns.2006.08.025. PMID 17210334
- [Background] Lin CY, Cheng PH, Fang SY. Mucosal changes in rhinitis medicamentosa. Ann Otol Rhinol Laryngol. 2004 Feb;113(2):147-51. doi: 10.1177/000348940411300213. PMID 14994772
- [Background] Cam B, Sari M, Midi A, Gergin O. Xylitol treats nasal mucosa in rhinitis medicamentosa: an experimental rat model study. Eur Arch Otorhinolaryngol. 2019 Nov;276(11):3123-3130. doi: 10.1007/s00405-019-05605-3. Epub 2019 Aug 29. PMID 31468129
- [Background] Suh SH, Chon KM, Min YG, Jeong CH, Hong SH. Effects of topical nasal decongestants on histology of nasal respiratory mucosa in rabbits. Acta Otolaryngol. 1995 Sep;115(5):664-71. doi: 10.3109/00016489509139384. PMID 8928640
- [Background] Tas A, Yagiz R, Yalcin O, Uzun C, Huseyinova G, Adali MK, Karasalihoglu AR. Use of mometasone furoate aqueous nasal spray in the treatment of rhinitis medicamentosa: an experimental study. Otolaryngol Head Neck Surg. 2005 Apr;132(4):608-12. doi: 10.1016/j.otohns.2005.01.010. PMID 15806055
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Tait SD, Kallogjeri D, Chidambaram S, Schneider J, Piccirillo JF. Psychometric and Clinimetric Validity of the Modified 25-Item Sino-Nasal Outcome Test. Am J Rhinol Allergy. 2019 Sep;33(5):577-585. doi: 10.1177/1945892419851622. Epub 2019 May 28. No abstract available. PMID 31134810
- [Background] Hopkins C, Gillett S, Slack R, Lund VJ, Browne JP. Psychometric validity of the 22-item Sinonasal Outcome Test. Clin Otolaryngol. 2009 Oct;34(5):447-54. doi: 10.1111/j.1749-4486.2009.01995.x. PMID 19793277
- [Background] Lipan MJ, Most SP. Development of a severity classification system for subjective nasal obstruction. JAMA Facial Plast Surg. 2013 Sep-Oct;15(5):358-61. doi: 10.1001/jamafacial.2013.344. PMID 23846399
- [Background] Taverner D, Bickford L, Shakib S, Tonkin A. Evaluation of the dose-response relationship for intra-nasal oxymetazoline hydrochloride in normal adults. Eur J Clin Pharmacol. 1999 Sep;55(7):509-13. doi: 10.1007/s002280050665. PMID 10501820
- [Background] Akerlund A, Klint T, Olen L, Rundcrantz H. Nasal decongestant effect of oxymetazoline in the common cold: an objective dose-response study in 106 patients. J Laryngol Otol. 1989 Aug;103(8):743-6. doi: 10.1017/s0022215100109958. PMID 2671220
- [Background] Druce HM, Ramsey DL, Karnati S, Carr AN. Topical nasal decongestant oxymetazoline (0.05%) provides relief of nasal symptoms for 12 hours. Rhinology. 2018 Dec 1;56(4):343-350. doi: 10.4193/Rhin17.150. PMID 29785414
- [Background] Saratziotis A, Emanuelli E, Zanotti C, Mireas G, Pavlidis P, Ferfeli M, Hajiioannou J. Endoscopic sinus surgery outcomes in CRS: quality of life and correlations with NOSE scale in a prospective cohort study. Eur Arch Otorhinolaryngol. 2021 Apr;278(4):1059-1066. doi: 10.1007/s00405-020-06334-8. Epub 2020 Sep 8. PMID 32897442
- [Background] Kandathil CK, Saltychev M, Abdelwahab M, Spataro EA, Moubayed SP, Most SP. Minimal Clinically Important Difference of the Standardized Cosmesis and Health Nasal Outcomes Survey. Aesthet Surg J. 2019 Jul 12;39(8):837-840. doi: 10.1093/asj/sjz070. PMID 30873533
- [Background] Baroody FM, Brown D, Gavanescu L, DeTineo M, Naclerio RM. Oxymetazoline adds to the effectiveness of fluticasone furoate in the treatment of perennial allergic rhinitis. J Allergy Clin Immunol. 2011 Apr;127(4):927-34. doi: 10.1016/j.jaci.2011.01.037. Epub 2011 Mar 5. PMID 21377716